CLINICAL TRIAL: NCT06594731
Title: Belt Squat Training for Individuals with Chronic Non-Specific Low Back Pain - a Feasibility Study
Brief Title: Belt Squat Training for Non-Specific Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mathias Kristiansen (Other)
Collaborators: Aalborg University Hospital (Other)
Responsible Party: Sponsor-Investigator, Mathias Kristiansen, Associate Professor, Aalborg University
Organization: Aalborg University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: N-20230063
Record Dates: First submitted 2024-09-03; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Low Back Pain
Keywords: Feasibility study
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Low back pain patients (Experimental): Low back pain subjects performing hip belt squat training twice per week for 6 weeks.
  Interventions: Other: Hip belt squat training
- Healthy individuals (Active Comparator): Healthy individuals performing hip belt squat training twice per week for 6 weeks.
  Interventions: Other: Hip belt squat training

INTERVENTIONS:
Other: Hip belt squat training — Hip belt squat training performed twice per week for 6 weeks

SUMMARY:
The purpose of this project is to investigate the feasibility of using belt squat as an exercise intervention for people with chronic low back pain. We will recruit people with chronic low back pain as well as asymptomatic controls

DETAILED DESCRIPTION:
The purpose of the current project is to evaluate the feasibility of performing belt squats in healthy participants and persistent non-specific low back pain (LBP) patients.

For this project we wish to recruit 20 healthy volunteers 20 volunteers LBP patients through notices at Aalborg University, on www.forsog.dk, and on Facebook. The following inclusion and exclusion criteria will be used for the healthy subjects:

Healthy men and women, age 18-60.

And for the LBP patients:

Non-specific LBP for more than twelve weeks without major sciatica (back pain >leg pain), age 18-60.

Exclusion criteria pertinent to all subjects were:

Leg pain greater than back pain, neuromuscular disorders, spinal or lower extremity fractures, infections, cancer, osteoporosis, dementia, BMI>35, current substance abuse, former lumbar surgery, persistent pain syndromes other than back pain, inflammatory rheumatic diseases.

In the study, participants will perform hip belt squat training twice per week for 6 weeks.

To test the feasibility of performing hip belt squat training in healthy participants and persistent LBP patients the project will be based on the Bowen feasibility model. This model lists eight different focus areas for feasibility studies, where this particular sub-project will focus on four of these areas being: acceptability, demand, implementation, and practicality.

To test the acceptability and demand, subjects will be interviewed on their satisfaction, intention to continue use, actual use, perceived appropriateness, and perceived demand of the training.

Implementation and practicality will be assessed by evaluation of the degree of execution, success or failure of execution, factors affecting implementation ease or difficulty, positive/negative effects on participants, ability of participants to carry out the training activities and a cost analysis.

Lastly, to test the acceptance of methods relevant to the training, measures on lumbar flexibility, muscle strength, muscle mass (DEXA scan), pain sensitivity (pressure-pain threshold, PPT) using a handheld pressure algometer (Somedic, Sweden), muscle activity (Electromyographic measurement, EMG) and the following questionnaires: Fear-avoidance Beliefs Questionnaire (FABQ), Oswestry Disability Index (ODI) (which ranges from 0 (no disability) to 100 (bedridden)), health-related quality of life as measured by EuroQOL-5D (EQ-5D) (ranging from -0.596 to 1, with higher scores indicating better quality of life) will be carried out

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women
* Men and women with non-specific low back pain for more than twelve weeks

Exclusion Criteria:

* Leg pain greater than back pain
* Neuromuscular disorders
* Spinal or lower extremity fractures
* Infections
* Cancer
* Osteoporosis
* Dementia
* Current substance abuse
* Former lumbar surgery
* Persistent pain syndromes other than back pain
* Inflammatory rheumatic diseases

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-06-15 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Acceptability | Immediately after the intervention
  Acceptability of the intervention will be assessed using a 5 point likert scale ranging from completely agree to completely disagree on whether the intervention was acceptable or not.
Demand | Immediately after the intervention
  Demand of the intervention will be assessed using a 5 point likert scale ranging from completely agree to completely disagree on whether the participants wish to incorporate belt squats into their future training.
Implementation | Immediately after the intervention
  Implementation of the intervention will be assessed using a 5 point likert scale ranging from completely agree to completely disagree on whether the intervention was feasible or not.
Practicality | Immediately after the intervention
  Practicality will be assessed by evaluation of the adherence level, computed as the percentage of completed training sessions.

SECONDARY OUTCOMES:
Pain sensitivity | Assessed at baseline and immediately after the intervention period
  Pressure-pain threshold was assessed using a handheld pressure algometer.
Muscle strength | Assessed at baseline and immediately after the intervention period
  Muscle strength was assessed in the hop belt squat exercise using a 5 repetition maximum test
Lumbar flexibility | Assessed at baseline and immediately after the intervention period
  Lumbar flexibility was assessed using a custom made test.
Muscle activity | Assessed at baseline and immediately after the intervention period
  Electromyography was used to assess muscle activation.
Oswetry Disability index | Assessed at baseline and immediately after the intervention period
  A questionnaire measuring the degree of disability, which ranges from 0 (no disability) to 100 (bedridden).
Health related quality of life | Assessed at baseline and immediately after the intervention period
  A questionnaire measuring the easured health-related quality of life (EuroQOL-5D), ranging from -0.596 to 1, with higher scores indicating better quality of life.
Fear-avoidance Beliefs Questionnaire | Assessed at baseline and immediately after the intervention period
  Fear-avoidance Beliefs Questionnaire (FABQ) measuring the amount of kinesiophobia, ranging from 0-96 with higher scores indicating higher levels of fear avoidance belief.
Body composition | Assessed at baseline and immediately after the intervention period
  To assess changes in body composition a DEXA scan was performed. This test quantified lean body mass (kg) and fat mass (kg).

CONTACTS AND LOCATIONS:
Locations (1):
- Aalborg University, Gistrup, Denmark

IPD SHARING:
Plan to Share IPD: No